CLINICAL TRIAL: NCT00250185
Title: The Role of Nitrite in Preconditioning Mediated Tolerance to Ischemic Stress
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 060024; 06-H-0024
Record Dates: First submitted 2005-11-05; First posted 2005-11-07 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2008-08-22

CONDITIONS: Ischemic Stress; Transient Non-Lethal Ischemia
Keywords: Ischemia Tolerance; Endothelial Function; Forearm Blood Flow; Muscle Recovery; Inflammation; Healthy Volunteer; HV
MeSH Terms: conditions — Inflammation | interventions — sodium nitrate; Acetylcholine

INTERVENTIONS:
Drug: Sodium Nitrate
Drug: Acetylcholine

SUMMARY:
Many studies have shown that if the human body is stressed by a lack of blood flow for a short period of time, the body develops defenses to make the body more resistant to a future stress from lack of blood flow. This natural defense system is called preconditioning. Finding medications that have a preconditioning effect to protect against damage from loss of blood flow would be of great help in the treatment of diseases such as heart attacks and stroke that occur because of blockages of blood flow.

Predicting future heart attacks or strokes is very difficult and makes it difficult to study medications that could have a preconditioning effect. However, it has recently been recognized that we can mimic the preconditioning effect in the human arm, by blocking blood flow using a blood pressure cuff under pressure. Here, blowing up the cuff for 5 minutes and then letting the pressure out for 5 minutes and repeating this process twice more (a way to precondition the arm), has been shown to improve blood vessel function in response to a longer period of blood pressure cuff inflation (20 minutes).

As nitrite, a naturally occurring blood substance, has biological effects suggesting that it may mimic preconditioning. The main objective of this study is to assess whether nitrite is equivalent to preconditioning in its capacity to protect the forearm blood flow in response to a 20 minute blockage of blood flow by blood pressure cuff inflation of the forearm.

We hypothesize that in human subjects the ischemic preconditioning program works through activation of the pool of nitrite in the blood stream. Moreover, we propose that nitrite treatment will improve (1) blood vessel recovery (2) skeletal muscle blood flow and (3) skeletal muscle mitochondrial function and (4) reduce the activation of inflammation in response to the 20 minute stress of blood pressure cuff inflation.

DETAILED DESCRIPTION:
Many studies have shown that if the human body is stressed by a lack of blood flow for a short period of time, the body develops defenses to make the body more resistant to a future stress from lack of blood flow. This natural defense system is called preconditioning. Finding medications that have a preconditioning effect to protect against damage from loss of blood flow would be of great help in the treatment of diseases such as heart attacks and stroke that occur because of blockages of blood flow.

Predicting future heart attacks or strokes is very difficult and makes it difficult to study medications that could have a preconditioning effect. However, it has recently been recognized that we can mimic the preconditioning effect in the human arm, by blocking blood flow using a blood pressure cuff under pressure. Here, blowing up the cuff for 5 minutes and then letting the pressure out for 5 minutes and repeating this process twice more (a way to precondition the arm), has been shown to improve blood vessel function in response to a longer period of blood pressure cuff inflation (20 minutes).

As nitrite, a naturally occurring blood substance, has biological effects suggesting that it may mimic preconditioning. The main objective of this study is to assess whether nitrite is equivalent to preconditioning in its capacity to protect the forearm blood flow in response to a 20 minute blockage of blood flow by blood pressure cuff inflation of the forearm.

We hypothesize that in human subjects the ischemic preconditioning program works through activation of the pool of nitrite in the blood stream. Moreover, we propose that nitrite treatment will improve (1) blood vessel recovery (2) skeletal muscle blood flow and (3) skeletal muscle mitochondrial function and (4) reduce the activation of inflammation in response to the 20 minute stress of blood pressure cuff inflation.

ELIGIBILITY:
* INCLUSION CRITERIA:

Subjects must be 18-45 years of age.

Subject must be in good health.

Subjects must provide informed, written consent for participation in this study.

Female subjects of childbearing age must have a negative pregnancy test.

EXCLUSION CRITERIA:

Subjects with a history of cardiac, pulmonary, peripheral vascular, or mitochondrial disease or diabetes mellitus.

Subjects with a history or evidence of present or past hypertension (blood pressure greater than 140/90 mmHg), hypercholesterolemia (LDL cholesterol greater than 160 mg/dL).

Subjects with abnormal EKG other than sinus bradycardia.

Subjects who have a history of smoking within three months.

Subjects with anemia (defined as hemoglobin less than 9 g/dL).

BMI greater than 30.

Subjects with a history of reaction to a medication or other substance characterized by dyspnea and cyanosis will not participate in this study.

Subjects with G6PD deficiency.

Subjects with a baseline methemoglobin level greater than 1.5%.

Lactating females who are breastfeeding, will not participate since nitrite crosses into breast milk and could cause methemoglobinemia in the infant.

No volunteer subject will be allowed to take any prescription medication (oral contraceptive agents are allowed). Vitamin supplements, herbal preparations, nutriceuticals or other 'alternative therapies' must be stopped for two weeks prior to study and aspirin, tylenol and NSAIDs must also be discontinued two weeks prior to study.

Subjects with a blood pressure of less than 90/60 mmHg or mean arterial pressure (MAP) less than 70 mmHg on the study day will be excluded from the protocol.

Positive for HIV or hepatitis A or B or positive for syphilis.

Subjects with a history of placement or insertion of any metal devices including pacemakers, cardiac defibrillators, cochlear implants, aneurysm clips, neural stimulators, insulin pumps or foreign bodies, such as, metal shavings will be excluded from participation in the MRS.

Subjects with a history of claustrophobia or an inability to lie on their backs will be excluded from the MRS sub-study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 135
Dates: Start 2005-11-01; Primary Completion 2007-06-09 (Actual); Study Completion 2007-06-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Dawn B, Bolli R. Role of nitric oxide in myocardial preconditioning. Ann N Y Acad Sci. 2002 May;962:18-41. doi: 10.1111/j.1749-6632.2002.tb04053.x. PMID 12076960
- [Background] Gladwin MT, Shelhamer JH, Schechter AN, Pease-Fye ME, Waclawiw MA, Panza JA, Ognibene FP, Cannon RO 3rd. Role of circulating nitrite and S-nitrosohemoglobin in the regulation of regional blood flow in humans. Proc Natl Acad Sci U S A. 2000 Oct 10;97(21):11482-7. doi: 10.1073/pnas.97.21.11482. PMID 11027349
- [Background] Zweier JL, Wang P, Samouilov A, Kuppusamy P. Enzyme-independent formation of nitric oxide in biological tissues. Nat Med. 1995 Aug;1(8):804-9. doi: 10.1038/nm0895-804. PMID 7585184